CLINICAL TRIAL: NCT07319741
Title: Clinical and Radiographic Evaluation of Single Visit Pulpectomy in Primary Molars for (5-7) Years Old Children Using Rotary and Manual Instrumentation: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Outcomes of Rotary Instrumentation in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anfal mohamed elmotaz almogtaba (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Anfal mohamed elmotaz almogtaba, Master's student, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rotary Files in Children
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Pulpectomy; Irreversible Pulpitis
Keywords: Single visit pulpectomy; Rotary Instrumentation; Manual Instrumentation; Pain; swelling; radiographic outcomes
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study will include two groups with an allocation ratio of 1:1.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The co-supervisor and main supervisor will also be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Single-Visit Pulpectomy using Rotary instrumentation (Active Comparator): This group will include patients with irreversible pulpitis who will undergo single-visit pulpectomy using rotary instrumentation
  Interventions: Procedure: Rotary Instrumentation
- Group2: Single-visit pulpectomy using manual instrumentation (Active Comparator): This group will include patients with irreversible pulpitis who will undergo single-visit pulpectomy using manual instrumentation
  Interventions: Procedure: Manual Instrumentation

INTERVENTIONS:
Procedure: Rotary Instrumentation — Single visit pulpectomy using rotary instrumentation
  Arms: Group 1: Single-Visit Pulpectomy using Rotary instrumentation
Procedure: Manual Instrumentation — Single visit pulpectomy using manual instrumentation
  Arms: Group2: Single-visit pulpectomy using manual instrumentation

SUMMARY:
This study will evaluate the clinical and radiographic outcomes of rotary versus manual pulpectomy in children with irreversible pulpitis.A single-visit pulpectomy will be performed for all patients. Participants will be allocated to rotary instrumentation using Fanta AF Baby files or manual step-back instrumentation with K-files. Canals will be irrigated with 17% EDTA and 1% sodium hypochlorite, obturated with Metapex, and restored with glass ionomer cement and stainless-steel crowns. Primary outcomes will assess clinical success at 3, 6, 9, and 12 months, while secondary outcomes will evaluate postoperative pain and radiographic success at 6 and 12 months.

DETAILED DESCRIPTION:
In this study, the principal investigator will screen participants to ensure eligibility and obtain comprehensive medical and dental histories from their parents or legal guardians, along with informed consent. All participants will undergo thorough clinical and radiographic examinations to confirm a diagnosis of irreversible pulpitis and suitability for pulpectomy. Local anesthesia will be administered, followed by caries removal, access cavity preparation, and pulpal extirpation. Working length will be determined radiographically, and participants will be allocated into two groups based on instrumentation technique: Group 1 will receive rotary instrumentation using Fanta AF Baby files with a crown-down approach, while Group 2 will undergo manual instrumentation using K-files with a step-back technique. Irrigation will involve 17% EDTA gel and 1% sodium hypochlorite, and canals will be obturated with Metapex, followed by restoration with glass ionomer cement and stainless-steel crowns in the same visit. The primary outcome will assess clinical success at 3, 6, 9, and 12 months post-treatment, defined by the absence of soft tissue swelling, tenderness, sinus tract, fistula, or pathological mobility. Secondary outcomes will include evaluation of postoperative pain intensity using a modified Wong-Baker Pain Rating Scale and radiographic success at 6 and 12 months, defined by the absence of root resorption, periodontal ligament widening, or periapical/furcal radiolucency.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-7 years with irreversible pulpitis of primary molars.
* History of spontaneous pain with a deep carious lesion.
* Parents who approve to write informed consent.

Exclusion Criteria:

* Medically compromised children.
* Children with a history of allergic reaction to the materials used in the study.
* Children with non-restorable teeth.
* Teeth with resorbed roots (more than two-thirds of root length).
* Extensive internal or external root resorption visible in periapical Radiographs.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Clinical success of Pulpectomy procedure | 12 months
  The primary outcome of this study will be the assessment of clinical success of the both instrumentation techniques (Manual and Rotary instrumentation), evaluated at 3, 6, 9, and 12 months post-treatment. Clinical success will be defined based on binary assessment by the absence of soft tissue swelling, tenderness to percussion (Performed by the back of the mirror), sinus tract, fistula, and pathologic mobility

SECONDARY OUTCOMES:
Evaluation of Radiographic Success of Pulpectomy | 12 months
  Another secondary outcome of this study will be the radiographic evaluation of treatment after manual and rotary instrumentation based on binary assessment at 6 and 12 months postoperatively. Radiographic success will be defined as the absence of internal or external root resorption, loss of lamina dura integrity, periodontal ligament widening, or alveolar bone resorption in the periapical region. The presence of any of these findings or periapical/furcal radiolucency will be considered radiographic failure.
  13. Participant Timeline

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided